CLINICAL TRIAL: NCT07321366
Title: Efficacy and Tolerability of Cryoneurolysis Treatment in Disabling and/or Painful Hypertonia of the Shoulder and Elbow in Patients With Cerebral Palsy Who Have Reached a Therapeutic Impasse a Pilot Study
Brief Title: Pilot Study on the Efficacy and Tolerability of Cryoneurolysis Treatment in Disabling and/or Painful Hypertonia of the Shoulder and Elbow in Patients With Cerebral Palsy
Acronym: OP-CRYO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Médico-Chirurgical de Réadaptation des Massues Croix Rouge Française (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025_06_OPCRYO_DM; 2025-A01180-49 (Other: ANSM)
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cryoneurolise treatment (Experimental): After testing the function following treatment with a motor block, the patient receives an indication for cryoneurolysis treatment.
  Interventions: Procedure: Cryoneurlysis

INTERVENTIONS:
Procedure: Cryoneurlysis — Ultrasound-guided percutaneous cryoneurolysis (CN) is a new, minimally invasive approach that allows the treatment of hypertonia by reversibly blocking nerve conduction secondary to axonotmesis. Although this approach has shown promising results with real benefits in the management of spasticity, its efficacy has not been determined in CP. CN therefore represents a therapeutic alternative between toxin injections and radical surgery in the management of complex tone disorders in CP, for achieving individualised objectives, including pain relief.

SUMMARY:
The main objective of this study is to evaluate the achievement of personalised short- and medium-term objectives of this selective treatment of hypertonia by ultrasound-guided perineural percutaneous cryoneurolysis at the shoulder and elbow, in a population of patients with cerebral palsy with spastic, dyskinetic or dyskinetic, or mixed disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cerebral palsy treated at the CMCR des Massues, regardless of their functional status as defined by their gross motor function level on the GMFCS (Gross Motor Function Classification System) and their manual ability level on the MACS (Manual Ability Classification System).
* Presenting with disabling and/or painful muscle hyperactivity in the shoulder and/or elbow,
* Aged over 12 years,
* At a therapeutic impasse: contraindicated or refusing surgery, contraindication or insufficient efficacy of oral treatments (analgesics, baclofen, Artane), too short duration of efficacy of toxin injections (<3 months) and/or dose-weight limitation not allowing treatment of all necessary sites.
* Patient (and legal representatives in the case of a minor patient or guardian/curator in the case of an adult patient under legal protection measures) who has been informed and has signed the informed consent form for participation in the research,
* Patient affiliated with a social security scheme.

Exclusion Criteria:

* - Patients who have received a botulinum toxin injection (any location) within 3 months prior to inclusion.
* Change in analgesic and/or antispastic treatment within 5 weeks prior to inclusion - Refusal to allow the patient's medical data to be used for research purposes
* Contraindication to peripheral motor block and/or cryoneurolysis (haemostasis disorder, skin infection, Raynaud's syndrome, cryoglobulinaemia, cold urticaria).
* Pregnant/breastfeeding patients.
* Cognitive and/or behavioural disorders that prevent participation in the study or giving consent to participate

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Goal Assessment Scale | 1st visit, after cryoneurolysis treatment, 3 Months follow-up, 6 Months follow up, 9 Months follow-up, 12 Months follow-up
  Goal Assessment Scale is an individualized patient-centered outcome measure that quantifies the effects of an intervention based on personal goals. It involves collaboration among patients, caregivers, and healthcare professionals to identify and set meaningful treatment goals. GAS allows for the measurement of the extent to which these goals are met, providing a standardized approach to evaluate progress.

SECONDARY OUTCOMES:
Clinical tolerability | After cryoneurolysis treatment, 3 Months follow-up, 6 Months follow up, 9 Months follow-up, 12 Months follow-up
  The evaluation will be carried out, on the one hand, by quantifying the occurrence of adverse events following cryoneurolysis treatment. Once the effects have been confirmed, classification will be carried out by referring to the different grades of clinical classification on the NCI CTCAE version 5.0 scale (Common Terminology Criteria for Adverse Events).
Change in muscle structure | 1st visit, after cryoneurolysis treatment, 3 Months follow-up, 6 Months follow up, 9 Months follow-up, 12 Months follow-up
  The change in muscle structure of the muscles innervated by the cryoneurolysed nerve will be assessed using the modified Heckmatt scale. This scale allows for the evaluation of potential echogenic changes in spastic muscles (echogenicity), indicating the level of fibrotic change.
Muscle hyperactivity | 1st visit, after cryoneurolysis treatment, 3 Months follow-up, 6 Months follow up, 9 Months follow-up, 12 Months follow-up
  The modified Ashworth scale (19,20) will be used to quantify spasticity in patients who exhibit resistance to passive mobilisation (muscle hyperactivity). The average absolute variation in muscle response to stretching applied at given speeds will be assessed using the Modified Tardieu Scale (MTS).
Active range of motion | 1st visit, after cryoneurolysis treatment, 3 Months follow-up, 6 Months follow up, 9 Months follow-up, 12 Months follow-up
  Active range of motion (AROM) - movement of a joint performed entirely by the person doing the exercise - and passive range of motion (PROM) - movement applied to a joint solely by another person - in the shoulder and elbow will be measured using a goniometer.
Joint Pain | 1st visit, after cryoneurolysis treatment, 3 Months follow-up, 6 Months follow up, 9 Months follow-up, 12 Months follow-up
  To assess pain in relation to a specific location in the shoulder and/or elbow, several tools can be used.
  We will preferably use a visual analogue scale from 0 to 10 to assess We prefer to use the Visual Analogue Scale from 0 to 10 to assess the intensity of pain. According to this self-assessment scale, the patient requires pain management if VAS ≥ 4/10.
Average Patient Satisfaction | 1st visit, after cryoneurolysis treatment, 3 Months follow-up, 6 Months follow up, 9 Months follow-up, 12 Months follow-up
  The average patient satisfaction in relation to the overall sensation in the event of a change will be assessed using a visual analogue scale (VAS), presented vertically to the patient and/or their carer. This scale has two sides (depending on the patient's age and cognitive level), with one side illustrated by emoticons of different colours corresponding to a score of 0: not at all satisfied to 10: perfectly satisfied, and one side in the form of a graduated scale from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- CMCR des Massues, Lyon, Rhône, France